CLINICAL TRIAL: NCT01070641
Title: RCT of Carvedilol vs Variceal Band Ligation in the Primary Prophylaxis of Oesophageal Variceal Haemorrhage
Brief Title: RCT of Carvedilol Versus Variceal Band Ligation in the Primary Prophylaxis of Oesophageal Variceal Haemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Syed hasnain Ali Shah, Aga Khan University Hospital, Karachi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCT carvidalol vs EVBL
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Portal Hypertension
Keywords: CARVEDILOL; VARICEAL BAND LIGATION; PRIMARY PROPHYLAXIS
MeSH Terms: conditions — Hypertension, Portal | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carvedilol (Active Comparator): Each patient will receive Carvedilol 12.5mg QD
  Interventions: Drug: Carvedilol
- Esophageal Variceal Band Ligation (Active Comparator): Each patient will undergo for serial esophageal variceal band ligations after 3 weeks of last session till the eradication of varices
  Interventions: Procedure: Esophageal variceal band ligation

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 12.5mg QD
  Other Names: carvida
  Arms: Carvedilol
Procedure: Esophageal variceal band ligation — Each patient will undergo for variceal band ligation after 3 weeks till the eradication of varices
  Other Names: EVBL
  Arms: Esophageal Variceal Band Ligation

SUMMARY:
Aim To compare Carvedilol with variceal band ligation in the prevention of first variceal bleed.

End points of trial Primary: Variceal hemorrhage Secondary: Death

Study design

Randomised controlled clinical trial. Results analysed for the above end points on an intention-to-treat basis.

DETAILED DESCRIPTION:
Patients from the Gastroenterology section of the Aga Khan University, Karachi, with liver cirrhosis and on endoscopy having grade II, or larger oesophageal varices and who have not bled previously from varices.

Method All suitable patients will be recruited after informed consent is given. Randomisation of treatment is by sealed envelopes prepared in batches of 20.

Carvedilol This will be administered as a once daily dose of 12.5mg.

Variceal band ligation Endoscopy will be performed ever two weeks until eradication of oesophageal varices. Eradication is achieved when no varices or only grade I varices (varices which are small and flatten on air insufflations in the oesophagus) are present. Subsequent endoscopy sessions will be progressively less frequent, at intervals of 3 months, 6 months and 12 months thereafter. Should varices recur, the protocol for eradication as described above will be re-instituted.

Follow-up This will take place in a dedicated clinic. First visit is six weeks after initiation of treatment and three monthly thereafter. Clinical and laboratory parameters will be obtained at each visit. All patients with alcoholic liver disease will be asked to provide an up-to-date status on drinking. Treatment will cease upon reaching any of these end-points: variceal haemorrhage, death or liver transplantation. Duration of follow-up is defined as time from randomisation to the above end points or to the last follow-up date available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis and on endoscopy having grade II, or larger oesophageal varices and who have not bled previously from varices.

Exclusion Criteria:

* Age <18 or > 75 years.
* Pregnant or lactating patients: patients of childbearing age who are not on contraception.
* Allergy to Carvedilol.
* Already on beta blockers or nitrates.
* Presence of malignancy that will significantly affect survival.
* Presence of severe systemic illness e.g. cardiorespiratory, active sepsis.
* Psychiatric disease or learning difficulty that will prevent the granting of informed consent.
* Presence of obstructive airways disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2002-06; Primary Completion 2011-02 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Variceal hemorrhage | one year

SECONDARY OUTCOMES:
death | one year

CONTACTS AND LOCATIONS:
Overall Officials: Syed hasnain A Shah, MBBS, FRCP, Principal Investigator — Aga Khan University Hospital, Karachi
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan